CLINICAL TRIAL: NCT03503474
Title: Combatting Bacterial Resistance in Europe - Clostridium Difficile Infections (COMBACTE-CDI, Understanding the Burden of Disease
Brief Title: COMBACTE-CDI Understanding the Burden of C. Difficile Infection
Acronym: COMBACTE-CDI
Status: Completed | Type: Observational
Sponsor: University of Leeds (Other)
Collaborators: Innovative Medicines Initiative (Other); UMC Utrecht (Other); Leiden University Medical Center (Other); National laboratory for Health, Environment and Food, Slovenia (Other); Universitätsklinikum Köln (Other); Universiteit Antwerpen (Other); National Institute for Infectious Diseases 'Lazzaro Sapllanzani', Italy (Other); Universität Tübingen (Other); Pfizer (Industry); GlaxoSmithKline (Industry); BioMérieux (Industry); AstraZeneca (Industry); Sanofi Pasteur, a Sanofi Company (Industry); Da Volterra (Industry)
Responsible Party: Principal Investigator, Professor Mark Wilcox, Brotherton Chair of Microbiology, University of Leeds
Other Study IDs: IRAS244784
Record Dates: First submitted 2018-04-11; First posted 2018-04-19 (Actual); Results first posted 2022-02-09 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-01

CONDITIONS: Clostridium Difficile Infection
MeSH Terms: conditions — Clostridium Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — residual diagnostic faecal samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CDI cases
  Interventions: Other: No intervention
- CDI negative controls
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — There is no intervention, this is observational only

SUMMARY:
Clostridium difficile infection (CDI) is the most common cause of antibiotic associated diarrhoea in the western world. The infection causes significant diarrhoea, which in some cases can be serious and lead to secondary complications and even death. The infection is particularly an issue in elderly, frail patient, who are often already burdened with several other medical issues. Recent work has demonstrated that numerous cases are missed, either due to inadequate diagnostic tests or lack of clinical suspicion.

The public-private partnership in COMBACTE-CDI will quantify the burden of CDI via a large, complex, multi-centre, multi-country study, and describe current management practices. An increased understanding of the CDI burden across Europe and better understanding of transmission of the organism will provide a basis for the further development of public health interventions and practices.

Based on a previous successful study model (EUCLID), hospitals/laboratories of interest which carry out diagnostic testing of samples from both in-patients and community patients (including Long-Term Care Facilities patients) will be approached for inclusion in the study. Samples sent to the sites on the selected study date (regardless of test requested) will be tested at a central laboratory for CDI to look for missed cases of CDI. A follow up case/control study will collect data on outcomes and risk factors. Data will be used to construct transmission models and cost effective-ness models. Ultimately, a best practice model for CDI management will be developed.

ELIGIBILITY:
Inclusion Criteria:

* Anyone who has a diarrhoeal faecal sample submitted to the laboratories in the study for testing on the day of interest, regardless of test requested

Exclusion Criteria:

* Any repeat samples

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Anyone who has a diarrhoeal faecal sample submitted to the laboratories in the study for testing on the day of interest, regardless of test requested
Sampling Method: Non-Probability Sample
Enrollment: 3240 (Actual)
Dates: Start 2018-06-11 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Wilcox, MD, Study Director — University of Leeds
Locations (1):
- University of Leeds, Leeds, West Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rupnik M, Viprey V, Janezic S, Tkalec V, Davis G, Sente B, Devos N, Muller BH, Santiago-Allexant E, Cleuziat P, Wilcox M, Davies K; COMBACTE-CDI consortium. Distribution of Clostridioides difficile ribotypes and sequence types across humans, animals and food in 13 European countries. Emerg Microbes Infect. 2024 Dec;13(1):2427804. doi: 10.1080/22221751.2024.2427804. Epub 2024 Nov 27. PMID 39535868

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Anyone who has a diarrhoeal faecal sample submitted to the laboratories in the study for testing on the day of interest, regardless of test requested. The result of this observational study did not impact on patient treatment and management at the submitting laboratories.
Pre-assignment Details: Residual samples received during the study period were tested for Clostridioides difficile infection (CDI) at the coordinating laboratory. Informed consent is not required for the use of anonymised residual material. The number of CDI cases and negative controls are the number of participants with a sample that returned a positive or negative test result, respectively. Duplicate samples were excluded and therefore not completed. Test result was not reported back to the laboratories.
Period: Overall Study
Arm/Group | CDI Cases | CDI Negative Controls
Started | 103 (The number of participant with a diarrhoeal sample that returned a positive test result at the coordinating laboratory. There is no intervention as this is an observational study only.) | 3050 (The number of participant with a diarrhoeal sample that returned a negative test result at the coordinating laboratory. There is no intervention as this is an observational study only.)
Completed | 103 | 3050
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: A clinical report form was requested 6 months after collection of residual diarrhoeal samples for all positive CDI cases and a proportion of CDI negative controls (case-control study analysis population). The number of baseline participants is different from the participant Flow module, and is the number of CDI cases with completed clinical report form and an appropriate number of CDI negative controls from the pool of samples received to obtain a ratio of approximately 1:4 (Cases:Controls)
Groups:
- Total: Total of all reporting groups
Arm/Group | CDI Cases | CDI Negative Controls | Total
Number analyzed (Participants) | 94 | 444 | 538
Age, Customized [Median (Inter-Quartile Range); unit: years] | 72 [51 to 81] | 55 [21 to 72] | 58 [28 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 203 | 254
  Male | 43 | 241 | 284
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 24 | 137 | 161
  Belgium | 0 | 13 | 13
  France | 3 | 24 | 27
  Greece | 1 | 4 | 5
  Ireland | 1 | 3 | 4
  Italy | 13 | 43 | 56
  Netherlands | 2 | 9 | 11
  Poland | 12 | 38 | 50
  Romania | 18 | 57 | 75
  Slovakia | 2 | 8 | 10
  Spain | 13 | 93 | 106
  Sweden | 5 | 15 | 20
Healthcare settings Hospital at time of sample collection [Count of Participants; unit: Participants] | 76 | 301 | 377
Healthcare settings Community at time of sample collection [Count of Participants; unit: Participants] | 18 | 143 | 161
Exposure to at least one antibiotic in the preceding 12 weeks to the sample [Count of Participants; unit: Participants] — Population: Number of participants with data on this study-specific baseline measure as reported in the clinical report form (data obtained 6 months after sample collection)
  Participants
    number analyzed (Participants) | 80 | 354 | 434
    (all) | 57 | 174 | 231
Contact with healthcare facilities in the preceding 6 months to the sample [Count of Participants; unit: Participants] — Population: Number of participants with data on this study-specific baseline measure as reported in the clinical report form (data obtained 6 months after sample collection)
  Participants
    number analyzed (Participants) | 80 | 372 | 452
    (all) | 60 | 183 | 243
Two or more co-morbidities [Count of Participants; unit: Participants] — Population: Number of participants with data on this study-specific baseline measure as reported in the clinical report form (data obtained 6 months after sample collection)
  Participants
    number analyzed (Participants) | 86 | 390 | 476
    (all) | 56 | 138 | 194
White cell count per microliter [Mean (Standard Deviation); unit: 10^9 cells/μL] — Population: Number of participants with data on this study-specific baseline measure as reported in the clinical report form (data obtained 6 months after sample collection)
  10^9 cells/μL
    number analyzed (Participants) | 70 | 291 | 361
    (all) | 14800 (13600) | 10300 (8000) | 11200 (9500)
Number of days of diarrhoea before the sample [Median (Inter-Quartile Range); unit: days] — Population: Number of participants with data on this study-specific baseline measure as reported in the clinical report form (data obtained 6 months after sample collection)
  days
    number analyzed (Participants) | 68 | 258 | 326
    (all) | 3 [1 to 7] | 3 [1 to 7] | 3 [1 to 7]
Number of recurrent (previous) CDI [Count of Participants; unit: Participants] — Population: Number of participants with data on this study-specific baseline measure as reported in the clinical report form (data obtained 6 months after sample collection)
  Participants
    number analyzed (Participants) | 82 | 444 | 526
    (all) | 6 | 0 | 6
Hospital admission within 30 days of sample [Count of Participants; unit: Participants] — A clinical report form was requested 6 months after collection of residual diarrhoeal samples for all positive CDI cases and a proportion of CDI negative controls (case-control study analysis population). Therefore all baseline characteristics presented were obtained retrospectively, including the information on whether the participant was admitted to hospital within 30 days after collection of that same sample, and is considered a study-specific measure. Population: Number of participants with data on this study-specific baseline measure as reported in the clinical report form (data obtained 6 months after sample collection)
  Participants
    number analyzed (Participants) | 87 | 408 | 495
    (all) | 13 | 43 | 56
30 days mortality rate [Count of Participants; unit: Participants] — A clinical report form was requested 6 months after collection of residual diarrhoeal samples for all positive CDI cases and a proportion of CDI negative controls (case-control study analysis population). Therefore all baseline characteristics presented were obtained retrospectively, including the information on whether the participant died within 30 days after collection of that same sample, and is considered a study-specific measure. Population: Number of participants with data on this study-specific baseline measure as reported in the clinical report form (data obtained 6 months after sample collection)
  Participants
    number analyzed (Participants) | 88 | 401 | 489
    (all) | 14 | 24 | 38

OUTCOME MEASURES:

1. Primary Outcome: The Number of Cases of CDI
Description: This outcome measure is to indicate the number of participants with a sample that returned a positive test result (=CDI cases) at the coordinating laboratory from the overall total number of participants. The number of CDI cases and negative controls are the number of participants with a sample that returned a positive or negative test result, respectively. Therefore the "CDI negative controls" arm did not return a positive test result. The proportion of participants that returned a positive test result compared to the total of participants (=number of participants in the "CDI cases" arm divided by the number of total participants in both arms) can be inferred from this outcome measure.
Time Frame: Samples were received between July and December 2018 (at time of diarrheal episode) and test performed during that timeframe to identify the number of CDI cases (positive test result) and the number of CDI negative controls (negative test result).
Population: The number of CDI cases and negative controls are the number of participants with a sample that returned a positive or negative test result, respectively. Therefore the "CDI negative controls" arms did not return a positive test result.
Measure: Count of Participants; unit: Participants
Arm/Group | CDI Cases | CDI Negative Controls
Number analyzed (Participants) | 103 | 3050
Participants | 103 | 0

ADVERSE EVENTS:
Time Frame: Mortality rate (within 30 days of sample collection) was reported 6 months after sample collection, and therefore did not impact on participant management and treatment. This is provided as a study-specific measure to report on the difference in 30 days mortality rate between CDI cases and CDI negative controls. The total number of participants at risk are the number of participants with data obtained on this study-specific measure, 6 months after sample collection.
Description: For this observational study, serious and other adverse events were not monitored/assessed as participants were not enrolled in a clinical trial. Therefore the number of participants at risk for serious and other adverse events is shown as "0". However, all cause mortality (within 30 days of sample) was reported as an observation only, to report on the difference in 30 days mortality rate between CDI cases and CDI negative controls
Arm/Group | CDI Cases | CDI Negative Controls
All-Cause Mortality (participants affected / at risk) | 14/88 | 24/401
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2018-04-17): https://cdn.clinicaltrials.gov/large-docs/74/NCT03503474/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-04): https://cdn.clinicaltrials.gov/large-docs/74/NCT03503474/SAP_001.pdf